CLINICAL TRIAL: NCT04747730
Title: Fostering Inmates' Well-being and Mental Health Through Transcendental Meditation: a Prison Pilot
Brief Title: Fostering Inmates' Well-being and Mental Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unfortunately, the trial couldn't take place as planned as the investigators didn't manage to recruit a sufficient number of participants.
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 251271
Record Dates: First submitted 2021-01-29; First posted 2021-02-10 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-01

CONDITIONS: Well-being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcendental Meditation training (Experimental): The intervention of the project is the teaching and learning of Transcendental Meditation technique. The technique involves the use of a sound (mantra) to effortlessly allow the mind to settle down to a state of inner calm. It is a simple, natural and effortless practise, and unlike other meditation strategies, it does not involve concentration or control of the mind. The practice does not require any religion, philosophy, or change in lifestyle. Once learned the technique, participants will practice it twice a day, 20 minutes every morning and 20 minutes in the afternoon.
  Interventions: Other: Transcendental Meditation training
- control (No Intervention): no intervention

INTERVENTIONS:
Other: Transcendental Meditation training — The programme targets inmates in HMP Warren Hill who are eligible to learn the meditation technique, who are staying in prison for at least six months since the beginning of the programme and who provide the signed informed consent. The sample of eligible inmates is approximately 190 inmates out of 250 currently in the prison. Inmates will be contacted by the research team in prison during introductory sessions of the research intervention.
  Arms: Transcendental Meditation training

SUMMARY:
The objective of the project was to provide an assessment of the impact of Transcendental Meditation on prison inmates' well-being. To achieve this goal the investigators conducted a before-and-after study in Her Majesty's Prison Warren Hill (HMP) (England). Meditation is correlated with better self-regulation and is innovative because it fosters generalisable psychological processes that support cognitive, emotional and behavioural regulation, with self-regulation being an important factor behind a variety of outcomes.

Unfortunately, the trial couldn't be completed as the investigators didn't manage to recruit a sufficient number of participants.

DETAILED DESCRIPTION:
The meditation intervention consists of teaching four one-hour lessons of the Transcendental meditation technique developed and offered by the David Lynch Foundation. The technique involves the use of a sound (mantra) to effortlessly allow the mind to settle down to a state of inner calm. Meditation enables those who have learned it and regularly practice it to be more self-aware and respond in a calmer and more considered manner to whatever happens in their present experience.

ELIGIBILITY:
Inclusion Criteria:

* any inmate with no history of drug or alcohol abuse
* recreational drug users who have refrained from using drugs for two weeks before learning the meditation technique
* alcohol or drug addicts who are recovering from alcohol or drug use and have refrained from drug use for at least three months before taking part to the programme

Exclusion Criteria:

* informed consent not signed.
* expected stay in HMP Warren Hill shorter than six months since the beginning of the project.
* drug users and alcoholics not in rehabilitation
* people with serious mental health problems
* people who do not speak English as a first language.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Mental health: - GHQ 12 - SF-12 Health survey | 4 months after training
  GHQ 12 was collected via survey questions.
  The General Health Questionnaire (GHQ) is a screening device for identifying minor psychiatric disorders in the general population and within community or non-psychiatric clinical settings such as primary care or general medical out-patients. Suitable for all ages from adolescent upwards - not children, it assesses the respondent's current state and asks if that differs from his or her usual state. It is therefore sensitive to short-term psychiatric disorders but not to long-standing attributes of the respondent.
Mental health: - GHQ 12 - SF-12 Health survey | 4 months after training
  SF-12 was collected via survey questions.
  The SF-12 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP).
Patience and trust | 4 months after training
  Two survey questions assessing propensity for delayed gratification:
  1. assessing propensity for delayed gratification using monetary values (scale 1 to 32, 32 is highest, 1 is lowest).
  2. assessing propensity for delayed gratification using subjective values (scale 0 to 10, higher numbers reflecting a greater propensity than lower ones).
  One survey question on trust: scale from 0 to 10 (0 is lowest, 10 is highest).
Positive reciprocity | 4 months after training
  Two survey questions:
  1. "When someone does me a favour are you willing to return it?" (scale from 0 to 10, where 0 is the lowest value and 10 the highest).
  2. Hypothetical scenario where someone helps the participant find their way. How much are they willing to provide as monetary reward for the help received? No scale. Outcome in pounds.

CONTACTS AND LOCATIONS:
Locations (1):
- HMP Warren Hill, Woodbridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No